CLINICAL TRIAL: NCT06755385
Title: Pilot Study on the Value of Bedside Pleuropulmonary Ultrasound in Patients With Sickle Cell Disease Presenting With Vaso-occlusive Crisis.
Acronym: DREPP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0347
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Pulmonary anomalies; Vaso-occlusive crisis; Acute chest syndrom; Pleuropulmonary ultrasound
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pleuropulmonary ultrasound — pleuropulmonary ultrasounds performed at D0, between D2 and D5 during hospitalization and at D-1 on discharge

SUMMARY:
Describe the proportion of patients with major sickle cell syndrome in vaso-occlusive crisis presenting at least one pleuropulmonary ultrasound abnormality during one of the ultrasounds performed at D0, between D2 and D5 during hospitalization and at D-1 of discharge.

We hypothesize that pleuropulmonary ultrasound will make it possible to detect the serious complications associated with vaso-occlusive crises in patients with major sickle cell syndrome earlier and more reliably, in departments where ultrasound tools are still underdeveloped, while avoiding the need for more conventional radiology examinations that cause radiation in multi-hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient agreeing to participate in the study
* Patient with sickle-cell disease consulted to the emergency department or hospitalized in a conventional internal medicine department for a clinical picture of severe vaso-occlusive crisis (CVO) requiring hospitalization.
* Hospitalization in the internal medicine department
* Possible re-inclusion in the event of a subsequent episode of severe CVO

Exclusion Criteria:

* Subject under guardianship or subject deprived of freedom.
* Primary acute chest syndrom (not following a crisis)
* Pulmonary pathologies interfering with pleuro-pulmonary echo analysis: pneumonectomy, pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sickle cell disease hospitalized in the internal medicine department of Grenoble University Hospital for vasoocclusive crisis.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Description of the proportion of patients with sickle cell disease in vasoocclusive crisis presenting at least one pleuropulmonary ultrasound abnormality at D0, between D2 and D5 during hospitalization and at D-1 of discharge. | 30 days
  Presence of abnormalities found during pleuropulmonary ultrasound scans performed in the medical department on D0, between D2 and D5 during hospitalization and on D-1 of discharge, in patients with major sickle cell syndrome presenting with vasoocclusive crisis, among the following:
  * Pulmonary condensations;
  * Pleural effusion: minimal, of moderate abundance (estimated volume < 500mL) or of great abundance (estimated volume > 500mL);
  * Confluent B lines (≥ 3 B lines per lung field).

SECONDARY OUTCOMES:
Evaluate the association between the ultrasound image and the clinical picture | 30 days
  Numbers and characteristics of abnormalities detected by EPP between D0, D2-J5 during hospitalization and D-1 of discharge, compared with numbers and characteristics of clinical abnormalities found between D0, D2-J5 during hospitalization and D-1 of discharge.
Evaluate the association between the ultrasound image detected and the occurrence of acute chest syndrom. | 30 days
  Number and characteristics of abnormalities detected by EPP between D0, D2-J5 during hospitalization and at D-1 of discharge, in patients progressing towards an acute chest syndrom, compared with the number and characteristics of abnormalities detected by EPP between D1 and D5 during hospitalization and at D-1 of discharge in patients not progressing towards an acute chest syndrom.
Evaluate the association between the ultrasound image detected and the severity of the acute chest syndrom | 30 days
  Numbers and characteristics of abnormalities detected by EPP between D1 and D5 during hospitalization and on D-1 of discharge, in relation to the severity of acute chest syndrom (oxygen demand, RF, transfer to ICU or intensive care unit).
Describe the evolution of abnormalities between visits at D0, between D2 and D5 (V1 and V2) during hospitalization and at D-1 of discharge, and their association with clinical evolution | 30 days
  Difference in proportion and characteristics of abnormalities detected by pleuropulmonary ultrasound on D0, between D2 and D5 (V1 and V2) during hospitalization and on D-1 of discharge.
Assess the prognostic value of discharge pleuropulmonary ultrasound in relation to re-hospitalization, occurrence of acute chest syndrom or early mortality (within 30 days) | 30 days
  Presence of at least one abnormality on day of discharge and number of re-hospitalizations, acute chest syndrom and 30-day mortality.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arlet JB. [Sickle cell disease imposes itself to French internists in the 21st century]. Rev Med Interne. 2023 Jul;44(7):325-327. doi: 10.1016/j.revmed.2023.05.006. Epub 2023 May 26. No abstract available. French. PMID 37246036
- [Background] Cheminet G, Mekontso-Dessap A, Pouchot J, Arlet JB. [Acute chest syndrome in adult sickle cell patients]. Rev Med Interne. 2022 Aug;43(8):470-478. doi: 10.1016/j.revmed.2022.04.019. Epub 2022 Jul 7. French. PMID 35810055
- [Background] Vichinsky EP, Neumayr LD, Earles AN, Williams R, Lennette ET, Dean D, Nickerson B, Orringer E, McKie V, Bellevue R, Daeschner C, Manci EA. Causes and outcomes of the acute chest syndrome in sickle cell disease. National Acute Chest Syndrome Study Group. N Engl J Med. 2000 Jun 22;342(25):1855-65. doi: 10.1056/NEJM200006223422502. PMID 10861320
- [Background] Castro O, Brambilla DJ, Thorington B, Reindorf CA, Scott RB, Gillette P, Vera JC, Levy PS. The acute chest syndrome in sickle cell disease: incidence and risk factors. The Cooperative Study of Sickle Cell Disease. Blood. 1994 Jul 15;84(2):643-9. PMID 7517723
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Bartolucci P, Habibi A, Khellaf M, Roudot-Thoraval F, Melica G, Lascaux AS, Moutereau S, Loric S, Wagner-Ballon O, Berkenou J, Santin A, Michel M, Renaud B, Levy Y, Galacteros F, Godeau B. Score Predicting Acute Chest Syndrome During Vaso-occlusive Crises in Adult Sickle-cell Disease Patients. EBioMedicine. 2016 Aug;10:305-11. doi: 10.1016/j.ebiom.2016.06.038. Epub 2016 Jun 29. PMID 27412264
- [Background] Lichtenstein D. Lung ultrasound in acute respiratory failure an introduction to the BLUE-protocol. Minerva Anestesiol. 2009 May;75(5):313-7. PMID 19412150
- [Background] Razazi K, Deux JF, de Prost N, Boissier F, Cuquemelle E, Galacteros F, Rahmouni A, Maitre B, Brun-Buisson C, Mekontso Dessap A. Bedside Lung Ultrasound During Acute Chest Syndrome in Sickle Cell Disease. Medicine (Baltimore). 2016 Feb;95(7):e2553. doi: 10.1097/MD.0000000000002553. PMID 26886600
- [Background] Koehl JL, Koyfman A, Hayes BD, Long B. High risk and low prevalence diseases: Acute chest syndrome in sickle cell disease. Am J Emerg Med. 2022 Aug;58:235-244. doi: 10.1016/j.ajem.2022.06.018. Epub 2022 Jun 11. PMID 35717760
- [Background] Colla JS, Kotini-Shah P, Soppet S, Chen YF, Molokie R, Prajapati P, Prendergast HM. Bedside ultrasound as a predictive tool for acute chest syndrome in sickle cell patients. Am J Emerg Med. 2018 Oct;36(10):1855-1861. doi: 10.1016/j.ajem.2018.07.006. Epub 2018 Jul 3. PMID 30017686
- [Background] Saah E, Lesnick BL. Lung Ultrasound in Sickle Cell: Sounds Like an Improvement in Acute Chest Diagnosis. Chest. 2023 Jun;163(6):1351-1352. doi: 10.1016/j.chest.2023.01.026. No abstract available. PMID 37295874
- [Background] Torres-Macho J, Aro T, Bruckner I, Cogliati C, Gilja OH, Gurghean A, Karlafti E, Krsek M, Monhart Z, Muller-Marbach A, Neves J, Sabio R, Serra C, Smallwood N, Tana C, Uyaroglu OA, Von Wowern F, Bosch FH; EFIM s ultrasound working group.. Point-of-care ultrasound in internal medicine: A position paper by the ultrasound working group of the European federation of internal medicine. Eur J Intern Med. 2020 Mar;73:67-71. doi: 10.1016/j.ejim.2019.11.016. Epub 2019 Dec 11. PMID 31836177